CLINICAL TRIAL: NCT00453063
Title: Placebo-Controlled Study of Mometasone Furoate Nasal Spray (MFNS) 200 mcg QD in the Treatment of Seasonal Allergic Rhinitis
Brief Title: Placebo-Controlled Study of Mometasone Furoate Nasal Spray (MFNS) 200 mcg Once Daily (QD) in the Treatment of Seasonal Allergic Rhinitis (Study P05067)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P05067
Record Dates: First submitted 2007-03-26; First posted 2007-03-28 (Estimated); Results first posted 2010-05-17 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MFNS 200 mcg QD (Experimental)
  Interventions: Drug: mometasone furoate
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: mometasone furoate — 50 mcg/spray, two sprays in each nostril once daily (ie, 200 mcg QD) in the morning
  Other Names: Nasonex; SCH 32088
  Arms: MFNS 200 mcg QD
Drug: Placebo — Two sprays in each nostril once daily in the morning
  Arms: Placebo

SUMMARY:
This study is designed to assess the effectiveness of mometasone furoate nasal spay (MFNS) once daily (QD) compared with placebo in subjects with seasonal allergic rhinitis (SAR) in reducing the total nasal symptom score and the total ocular symptom score.

ELIGIBILITY:
Inclusion Criteria:

* Must be 12 years of age or older, of either sex and of any race.
* Must have at least a 2-year documented history of SAR which exacerbates during the study season.
* Must have a positive skin-prick test response to an appropriate seasonal allergen at Screening (Visit 1). Immunoglobulin E (IgE)-mediated hypersensitivity to an appropriate seasonal allergen (ie, prevailing trees and/or grasses) must be documented by a positive response to the skin prick test with wheal diameter at least 3 mm larger than diluent control after 20 minutes.
* Must be clinically symptomatic at the Screening Visit.
* Must be clinically symptomatic at the Baseline Visit.
* Must be in general good health as confirmed by routine clinical and laboratory testing and electrocardiogram (ECG) results. Clinical laboratory test (complete blood count [CBC], blood chemistries, and urinalysis) must be within normal limits or clinically acceptable to the investigator and the sponsor.
* Must be free of any clinically significant disease, other than SAR, that would interfere with the study evaluations.

Exclusion Criteria:

* A history of anaphylaxis and/or other severe local reaction(s) to skin testing.
* A subject with asthma who requires chronic use of inhaled or systemic corticosteroids.
* Current or history of frequent, clinically significant sinusitis or chronic purulent postnasal drip.
* A subject with rhinitis medicamentosa.
* A history of allergies to more than two classes of medications or who are allergic to or cannot tolerate nasal sprays.
* A subject who has had an upper respiratory tract or sinus infection that required antibiotic therapy without at least a 14-day washout prior to the Screening Visit, or who has had a viral upper respiratory infection within 7 days before the Screening Visit.
* A subject who has nasal structural abnormalities, including large nasal polyps and marked septal deviations, which significantly interfere with nasal air flow.
* A subject who, in the opinion of the investigator, is dependent on nasal, oral, or ocular decongestants, nasal topical antihistamines, or nasal steroids.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 426 (Actual)
Dates: Start 2007-03; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

REFERENCES:
- [Result] Bielory L, Chun Y, Bielory BP, Canonica GW. Impact of mometasone furoate nasal spray on individual ocular symptoms of allergic rhinitis: a meta-analysis. Allergy. 2011 May;66(5):686-93. doi: 10.1111/j.1398-9995.2010.02543.x. Epub 2011 Jan 25. PMID 21261661

RESULTS

PARTICIPANT FLOW:
Groups:
- Mometasone Furoate Nasal Spray (MFNS): MFNS 200 mcg (two sprays in each nostril) once daily (QD) in the morning. Each spray is equal to 50 mcg.
- Placebo: Two sprays in each nostril once daily
Period: Overall Study
Arm/Group | Mometasone Furoate Nasal Spray (MFNS) | Placebo
Started | 211 | 215
Completed | 208 | 212
Not Completed | 3 | 3
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mometasone Furoate Nasal Spray (MFNS) | Placebo | Total
Number analyzed (Participants) | 211 | 215 | 426
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 18 | 30 | 48
  Between 18 and 65 years | 188 | 181 | 369
  >=65 years | 5 | 4 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140 | 130 | 270
  Male | 71 | 85 | 156

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Average AM Instantaneous (NOW) Total Nasal Symptom Score (TNSS) Averaged Over Days 2 to 15
Description: TNSS was defined as the sum of the following four nasal symptoms: rhinorrhea, nasal congestion/stuffiness, nasal itching, sneezing; each symptom scored on a scale of 0 = none, 1 = mild, 2 = moderate, and 3 = severe. The best possible score on this scale is 0 and the worst possible score on this scale is 12.
Time Frame: Baseline and 15 days
Population: All randomized participants were to be included in the analysis (intent-to-treat principle). However, subjects with a missing evaluation at a given visit or time point were not included in the analysis for that evaluation. This included participants without a baseline score for a given change-from-baseline evaluation.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mometasone Furoate Nasal Spray (MFNS) | Placebo
Number analyzed (Participants) | 209 | 213
units on a scale
  Baseline TNSS | 9.83 (1.56) | 9.69 (1.56)
  Change from Baseline in TNSS | -2.36 (2.07) | -1.71 (2.07)
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray (MFNS) vs Placebo; Test type: Superiority or Other; p = 0.001, ANCOVA

2. Primary Outcome: Change From Baseline in the Average AM Instantaneous (NOW) Total Ocular Symptom Score (TOSS) Averaged Over Days 2 to 15
Description: TOSS was defined as the sum of the following three ocular symptoms: redness of eyes, itching/burning eyes, and tearing/watering eyes; each symptom scored on a scale of 0 = none, 1 = mild, 2 = moderate, and 3 = severe. The best possible score on this scale is 0 and the worst possible score on this scale is 9.
Time Frame: Baseline and 15 days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mometasone Furoate Nasal Spray (MFNS) | Placebo
Number analyzed (Participants) | 209 | 213
units on a scale
  Baseline TOSS | 7.07 (1.54) | 7.01 (1.54)
  Change from Baseline in TOSS | -1.52 (1.59) | -1.36 (1.59)
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray (MFNS) vs Placebo; Test type: Superiority or Other; p = 0.304, ANCOVA

3. Secondary Outcome: Change From Baseline in AM NOW Nasal Congestion Score Averaged Over Days 2 to 15
Description: Nasal congestion was one of the symptoms measured in the TNSS and was scored on a scale of 0 = none, 1 = mild, 2 = moderate, and 3 = severe. The best possible score on this scale is 0 and the worst possible score on this scale is 3.
Time Frame: Baseline and 15 days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mometasone Furoate Nasal Spray (MFNS) | Placebo
Number analyzed (Participants) | 209 | 213
units on a scale
  Baseline Nasal Congestion Score | 2.66 (0.40) | 2.64 (0.40)
  Change from Baseline in Nasal Congestion Score | -0.54 (0.54) | -0.39 (0.54)
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray (MFNS) vs Placebo; Test type: Superiority or Other; p = 0.004, ANCOVA

4. Secondary Outcome: Change From Baseline in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Total Score at Endpoint (Last Post Baseline Evaluation Carried Forward)
Description: The RQLQ consisted of 28 items that fell into the following seven domains: activities, sleep, non-nose/eye symptoms, practical problems, nasal symptoms, eye symptoms, and emotional. Each of the items was scored from 0 = not troubled to 6 = extremely troubled, and the total of the seven domains was the primary focus of this quality of life evaluation. The best possible score on this scale is 0 and the worst possible score on this scale is 42. The Endpoint was the last post baseline evaluation carried forward and was Day 15 for the majority of the participants.
Time Frame: Baseline and 15 days
Population: The RQLQ tool is only validated in participants greater than or equal to 18 years of age, so it was only administered in this age group.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mometasone Furoate Nasal Spray (MFNS) | Placebo
Number analyzed (Participants) | 189 | 182
units on a scale
  Baseline RQLQ Total Score | 4.19 (0.97) | 4.42 (0.97)
  Change from Baseline in RQLQ Total Score | -1.63 (1.37) | -1.36 (1.37)
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray (MFNS) vs Placebo; Test type: Superiority or Other; p = 0.063, ANCOVA

5. Secondary Outcome: Change From Baseline in AM Peak Nasal Inspiratory Flow (PNIF) Averaged Over Days 2 to 15
Description: Participants were to measure nasal airflow twice daily (in the morning prior to study drug dosing and in the evening) using their PNIF meter. The highest of 3 assessments was to be recorded in the electronic diary. The PNIF meter limits were between 30 and 370 liters/minute. Normal values range between 100 and 150 liters/minute. A positive change from Baseline correlates with improved nasal air flow.
Time Frame: Baseline and 15 days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: liters/minute
Arm/Group | Mometasone Furoate Nasal Spray (MFNS) | Placebo
Number analyzed (Participants) | 209 | 213
liters/minute
  Baseline PNIF | 89.11 (37.2) | 88.85 (37.2)
  Change from Baseline in PNIF | 10.15 (21.1) | 8.24 (21.1)
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray (MFNS) vs Placebo; Test type: Superiority or Other; p = 0.356, ANCOVA

ADVERSE EVENTS:
Arm/Group | Mometasone Furoate Nasal Spray (MFNS) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/211 | 0/215
Other Adverse Events (participants affected / at risk) | 0/211 | 0/215

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the study.